CLINICAL TRIAL: NCT00502658
Title: Evaluation of Dietary Supplements (Shakes and Supplements) and Personal Energy Tracking Device to Promote and Maintain Healthy Weight
Brief Title: Dietary Supplements and Personal Energy Tracking Device to Promote and Maintain Healthy Weight
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pharmanex (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 007-001, WIRB 20070167
Record Dates: First submitted 2007-07-12; First posted 2007-07-17 (Estimated); Last update posted 2008-03-28 (Estimated); Status verified 2008-03

CONDITIONS: Overweight; Obesity
Keywords: Overweight; Obese; Dietary Supplements; Shakes; Nutrition; Overweight and Obese Adults (BMI 25-35)
MeSH Terms: conditions — Overweight; Obesity; Tremor | interventions — Minerals; Nutrients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Dietary supplement containing vitamins, minerals, and herbs
Behavioral: Shakes with nutrients and herbs
Behavioral: Control dietary supplement
Behavioral: Isocaloric, isonitrogenous control shakes without herbs
Behavioral: Personal energy tracking tool

SUMMARY:
Excessive body weight is becoming a concern around the world, for example over half of the American adult population is overweight or obese. The purpose of this study is to determine whether dietary supplements and shakes containing a combination of nutrients/ingredients individually shown in research studies to reduce hunger, enhance metabolism, reduce the body's ability to 'store' fat, and enhance energy, promote healthy body weight and composition over 12 weeks. A further study objective is to determine whether the inclusion of a personal, easy to use, energy tracking device for the measurement of daily energy intake and expenditure also helps with the promotion of healthy body weight and body composition.

In this prospective, blinded study 120 volunteers who meet the entrance criteria including a BMI 25-35 kg/m2 and sign the informed consent form to participate in a 12 week long study will be recruited. All subjects will consume a multi-vitamin, mineral and fish oil supplement. Subjects will be randomly assigned to a control or experimental group and stratified by BMI 25-30 and >30-35 kg/m2, age, and gender with an equal number of subjects in each strata across groups. A subset of subjects will also wear a personal energy tracking device. Subjects will be instructed how to incorporate the shakes and supplements into their current diet and encouraged to incorporate fruits, vegetables, whole grains, and other healthy foods into their current meals and to exercise at least 30 minutes five days per week.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-65 years of age.
* Body Mass Index (BMI) between 25-35
* Willing to stop taking any nutritional supplements

Exclusion Criteria:

* Currently taking weight loss medication or supplements
* Currently smoke
* Taking any prescription medications
* Experienced at least a 10 pound weight loss over the past 2 months.
* History of serious heart problems (i.e. heart attack, angina, bypass surgery).
* Diagnosed with diabetes (insulin or non-insulin dependent)
* Known history of gastrointestinal diseases (i.e. Crohn's disease, chronic diarrhea, Inflammatory Bowel Disease)
* Undergone surgical procedure for weight loss (i.e. gastroplasty, gastric by-pass, gastrectomy, stomach stapling, gastric banding, etc).
* History of stroke or seizure activity
* Medical conditions known to affect serum lipids
* History of uncontrolled hypertension or with a current measured blood pressure with diastolic above 90 or systolic above 140 mm Hg
* A total serum cholesterol above 240 mg/dL
* Known HIV infection
* Known history of depression and currently taking anti-depression medications
* Treated for cancer in the last 5 years
* Known allergies to supplements
* Known history of eating disorder (i.e. bulimia, anorexia nervosa)
* Known severe swallowing disorders
* For females, known to be pregnant or breast-feeding or trying to become pregnant
* Participating in another clinical (medical or nutritional) study or likely to be enrolled in another medical or nutritional protocol during this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2007-07; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Body weight changes | Several measurements over 12 weeks

SECONDARY OUTCOMES:
Biophotonic scanner score, blood chemistry and metabolic profiles, adverse events, subjects' supplement preference, quality of life measurements | Several measurements over 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Doug Burke, PhD, Principal Investigator — Pharmanex
Locations (1):
- Pharmanex, Provo, Utah, United States